CLINICAL TRIAL: NCT04124705
Title: A Multicenter, Randomized, Double-blind, Dose-conversion Study to Evaluate the Safety and Efficacy of Hormone Replacement Therapy With Armour® Thyroid Compared to Synthetic T4 (Levothyroxine) in Previously Hypothyroid Participants Who Are Euthyroid on T4 Replacement Therapy
Brief Title: A Study of Armour® Thyroid Compared to Synthetic T4 (Levothyroxine) in Previously Hypothyroid Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3014-201-002
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Results first posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Hypothyroidism; Thyroid Disease; Euthyroid; Thyroid Gland; Thyroid Hormones
MeSH Terms: conditions — Hypothyroidism; Thyroid Diseases | interventions — Thyroid (USP); Thyroxine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Armour® Thyroid (Experimental): Participants were randomized to receive Armour Thyroid at a dose corresponding to their pre-randomized dose of synthetic T4. During the first 18 to 36 weeks (titration period) the dose of Armour Thyroid could be titrated based on levels of thyroid stimulating hormone (TSH), in order to achieve TSH levels within the normal reference range (0.45 - 4.12 mIU/L, inclusive). Once TSH levels were within the normal reference range, participants continued to receive a stable dose of Armour Thyroid for an additional 12 weeks (stabilization period).
  Interventions: Drug: Armour® Thyroid
- Levothyroxine (Active Comparator): Participants were randomized to receive levothyroxine at their pre-randomized dose. During the first 18 to 36 weeks (titration period) the dose of levothyroxine could be titrated based on levels of TSH in order to achieve TSH levels within the normal reference range (0.45-4.12 mIU/L, inclusive). Once TSH levels were within the normal reference range, participants continued to receive a stable dose of levothyroxine for an additional 12 weeks (stabilization period).
  Interventions: Drug: Levothyroxine

INTERVENTIONS:
Drug: Armour® Thyroid — Administered orally once a day. the daily dose could range from 1/4 - 2 grains.
  Other Names: Desiccated thyroid extract; AGN-204771
  Arms: Armour® Thyroid
Drug: Levothyroxine — Administered orally once a day; the daily dose could range from 25- 200 µg.
  Other Names: Synthetic T4
  Arms: Levothyroxine

SUMMARY:
This study will evaluate the safe and effective dose conversion from levothyroxine (synthetic T4) therapy to Armour Thyroid therapy in participants who are on a stable dose of levothyroxine and have thyroid stimulating hormone (TSH) levels within the normal reference range.

DETAILED DESCRIPTION:
This study will include will include a Screening Period, double-blinded Titration Period (at least 18 weeks, up to 36 weeks), and a double-blinded Stabilization Period (12 weeks).

Participants will be randomized to receive either their same dose of levothyroxine or an approximately, matching dose of Armour Thyroid, using a dose-conversion chart based on the United States Pharmacopeia (USP) Drug Information 2000, which states that 1 grain of Armour Thyroid is equivalent to 100 mcg of levothyroxine.

During the Titration Period, Investigators will have the option to up-or down-titrate a participant's dose as needed based on the participant's TSH level (normal reference range 0.45 - 4.12 mIU/L, inclusive). At Week 18, if a participant's TSH levels are not within the normal reference range, the Investigator may up-or down-titrate the dose by continuing the Titration Period beyond Week 18 for up to a maximum of 3 additional titrations at 6-week intervals. Participants whose TSH levels have not normalized after the maximum 3 additional titrations will not enter the Stabilization Period.

At the end of the Titration Period, participants with TSH levels within normal reference range may enter the Stabilization Period. Depending on whether a participant requires additional dose titration after the Week 18 visit, the Stabilization Period may end at Week 30, 36, 42, or 48.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have a diagnosis of primary hypothyroidism made ≥ 12 months before study entry (Visit 1).
* Be on continuous thyroid replacement therapy with synthetic T4 for primary hypothyroidism for at least 12 months immediately prior to the Screening Visit (Visit 1).
* Be on a stable Food and Drug Administration (FDA)-approved daily dose of synthetic T4 for a minimum of 3 months prior to the Screening Visit (Visit 1). Must enter the study on the same stable dose.
* Have euthyroid status indicated by at least 1 documented TSH value within normal reference range (0.45 - 4.12 mIU/L, inclusive) at a minimum of 6 weeks and maximum of 12 months prior to the Screening Visit (Visit 1). Also have a confirmed TSH value within the normal reference range drawn at the Screening Visit (Visit 1).
* Male and female participants willing to minimize the risk of inducing pregnancy for the duration of the clinical study and follow-up period (35 days after last dose of study intervention).

Exclusion Criteria:

* Any clinical condition or previous surgery that might affect the absorption, distribution, biotransformation, or excretion of Armour Thyroid or synthetic T4.
* History of alcohol or other substance abuse within the previous 5 years.
* Known or suspected allergy or intolerance to any ingredients of Armour Thyroid, including its excipients, levothyroxine (T4), other thyroid replacement medications, or pork products.
* Have received active treatment with an investigational drug within 30 days or 5 half lives, whichever is longer, of Screening Visit (Visit 1).
* Current enrollment in an investigational drug or device study or participation in such a study within 60 days of entry into this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (28):
- United States (28):
  - Sponsor Site /ID# 237950, Birmingham, Alabama
  - Sponsor Site /ID# 237986, Little Rock, Arkansas
  - Sponsor Site /ID# 235210, Greenbrae, California
  - Sponsor Site /ID# 235716, Huntington Beach, California
  - Sponsor Site /ID# 238120, Sacramento, California
  - Sponsor Site /ID# 238026, Santa Clarita, California
  - Sponsor Site /ID# 238258, Van Nuys, California
  - Sponsor Site/ID# 235866, Denver, Colorado
  - Sponsor Site /ID# 235853, Fort Lauderdale, Florida
  - Sponsor Site /ID# 236809, West Palm Beach, Florida
  - Sponsor Site /ID# 235032, Atlanta, Georgia
  - Sponsor Site /ID# 237199, Columbus, Georgia
  - Sponsor Site /ID# 238088, Lawrenceville, Georgia
  - Sponsor Site /ID# 235714, Lexington, Kentucky
  - Sponsor Site /ID# 236701, Louisville, Kentucky
  - Sponsor Site /ID# 235202, Asheville, North Carolina
  - Sponsor Site/ID# 235204, Greenville, North Carolina
  - Sponsor Site /ID# 238023, Hickory, North Carolina
  - Sponsor Site /ID# 237137, Austin, Texas
  - Sponsor Site/ID# 238071, Austin, Texas
  - Sponsor Site/ID# 237652, Dallas, Texas
  - Sponsor Site/ID# 237655, Dallas, Texas
  - Sponsor Site /ID# 235870, El Paso, Texas
  - Sponsor Site /ID# 235860, Round Rock, Texas
  - Sponsor Site /ID# 235894, San Antonio, Texas
  - Sponsor Site /ID# 235211, Renton, Washington
  - Sponsor Site /ID# 236022, Spokane, Washington
  - Sponsor Site/ID# 236977, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled adults with a diagnosis of primary hypothyroidism who were taking a stable daily dose of synthetic T4 hormone (levothyroxine). Participants were enrolled at 27 sites in the United States.
Pre-assignment Details: Eligible participants were randomized equally to receive either their same dose of levothyroxine or a matching dose of Armour Thyroid at Baseline. The randomization was stratified by age (< 65 years, ≥ 65 years).
Period: Titration Period
Arm/Group | Armour® Thyroid | Levothyroxine
Started | 141 | 143
Received Study Treatment | 141 | 143
Completed | 115 | 124
Not Completed | 26 | 19
Not completed — Adverse Event | 9 | 5
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 1 | 1
Not completed — Lack of Efficacy | 2 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Non-compliance with Study Drug | 2 | 0
Not completed — Other | 4 | 9
Period: Stabilization Period
Arm/Group | Armour® Thyroid | Levothyroxine
Started | 115 | 124
Completed | 104 | 114
Not Completed | 11 | 10
Not completed — Adverse Event | 4 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of Efficacy | 4 | 2
Not completed — Protocol Deviation | 0 | 2
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Armour® Thyroid: Participants were randomized to receive Armour Thyroid at a dose corresponding to their pre-randomized dose of synthetic T4. During the first 18 to 36 weeks (titration period) the dose of Armour Thyroid could be titrated based on levels of TSH, in order to achieve TSH levels within the normal reference range (0.45 - 4.12 mIU/L, inclusive). Once TSH levels were within the normal reference range, participants continued to receive a stable dose of Armour Thyroid for an additional 12 weeks (stabilization period).
- Total: Total of all reporting groups
Arm/Group | Armour® Thyroid | Levothyroxine | Total
Number analyzed (Participants) | 141 | 143 | 284
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (12.94) | 53.4 (13.97) | 53.7 (13.45)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 108 | 109 | 217
  >= 65 years | 33 | 34 | 67
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 112 | 234
  Male | 19 | 31 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 21 | 38
  Not Hispanic or Latino | 124 | 122 | 246
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 14 | 10 | 24
  White | 124 | 124 | 248
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Thyroid Stimulating Hormone (TSH) Level [Mean (Standard Deviation); unit: mIU/L] | 1.81 (1.175) | 2.08 (1.507) | 1.95 (1.357)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Sustained TSH Response
Description: Sustained TSH response is defined as TSH values that are within the normal reference range of 0.45 to 4.12 mIU/L, inclusive, at both the end of Titration Period and the end of the Stabilization Period.
Time Frame: End of the titration period (Week 18, 24, 30, or 36) and end of the stabilization period (Week 30, 36, 42, or 48, depending on the length of the titration period).
Population: All randomized participants who took at least 1 dose of study intervention (intent-to-treat population). The non-responder imputation incorporating multiple imputation to handle missing data due to coronavirus disease 2019 (COVID-19) (NRI-C) was performed for participants who had missing TSH values either at the end of the Titration Period or at the end of the Stabilization Period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Armour® Thyroid | Levothyroxine
Number analyzed (Participants) | 141 | 143
percentage of participants | 60.76 [52.60 to 68.92] | 75.92 [68.65 to 83.19]
Statistical Analysis 1: Comparison: Armour® Thyroid vs Levothyroxine; The null hypothesis was that Armour Thyroid would be inferior to levothyroxine for the primary efficacy endpoint, sustained TSH response. The non-inferiority hypothesis test was performed at a 1-sided 2.5% level of significance (equivalent to a two-sided 5% level of significance); Test type: Non-Inferiority — If the lower limit of the 2-sided 95% confidence interval for stratified response rate difference was greater than the non-inferiority margin, the null hypothesis would be rejected and the noninferiority of Armour Thyroid to levothyroxine would be declared; Stratified Response Rate Difference = -15.16, 95% CI 2-sided [-26.10 to -4.23] — The response rate difference (Armour Thyroid group minus Levothyroxine group) and the 95% confidence interval were calculated using the Mantel-Haenszel-weighted method with the age group (age < 65 years or ≥ 65 years) as a stratification factor

2. Secondary Outcome: Percentage of Participants With a Titration TSH Response
Description: Titration TSH Response is defined as having a TSH value within the normal reference range of 0.45 to 4.12 mIU/L, inclusive, at the end of the Titration Period.
Time Frame: End of the titration period (Week 18, 24, 30, or 36)
Population: All randomized participants who took at least 1 dose of study intervention (intent-to-treat population). The non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was performed for participants who had missing TSH values at the end of Titration Period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Armour® Thyroid | Levothyroxine
Number analyzed (Participants) | 141 | 143
percentage of participants | 80.62 [74.05 to 87.18] | 91.13 [86.35 to 95.92]
Statistical Analysis 1: Comparison: Armour® Thyroid vs Levothyroxine; The null hypothesis was that Armour Thyroid would be inferior to levothyroxine for titration TSH response. The non-inferiority hypothesis test was performed at a 1-sided 2.5% level of significance; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Stratified Response Rate Difference = -10.52, 95% CI 2-sided [-18.65 to -2.38] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 35 days after last dose; maximum time on study was 48 weeks.
Arm/Group | Armour® Thyroid | Levothyroxine
All-Cause Mortality (participants affected / at risk) | 1/141 | 1/143
Serious Adverse Events (participants affected / at risk) | 4/141 | 7/143
Other Adverse Events (participants affected / at risk) | 15/141 | 9/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Armour® Thyroid (N=141) | Levothyroxine (N=143)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
OTITIS MEDIA (Infections and infestations) | 1 (1) | 0 (0)
PUNCTURE SITE ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 2 (2) | 0 (0)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
MIGRAINE WITH AURA (Nervous system disorders) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1) | 0 (0)
URETEROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1)
ADNEXA UTERI CYST (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Armour® Thyroid (N=141) | Levothyroxine (N=143)
FATIGUE (General disorders) | 7 (7) | 8 (8)
ANXIETY (Psychiatric disorders) | 8 (8) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/05/NCT04124705/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT04124705/SAP_001.pdf